CLINICAL TRIAL: NCT02498197
Title: Deltagerinvolverende Intervention Mod Fysiske Risikofaktorer for Muskel- og skeletbesvær i Byggebranchen
Brief Title: Participatory Intervention Among Construction Workers (IRMA11)
Acronym: IRMA11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Lars L. Andersen, Professor, PhD, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRMA11
Record Dates: First submitted 2015-06-29; First posted 2015-07-15 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participatory Intervention (Experimental): Participatory intervention with workers and their leaders. Workshops with presentation of work tasks with excessive physical load and subsequently plans to reduce these loads
  Interventions: Behavioral: Participatory Intervention
- Control (Active Comparator): Receive standard information about correct lifting technics, use of assistive technology, and ergonomics
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Participatory Intervention
  Arms: Participatory Intervention
Behavioral: Control
  Arms: Control

SUMMARY:
There is high prevalence of back pain and neck-shoulder pain among blue collar workers. Physical excessive exposures such as heavy lifting or working with a bended or twisted back are independent risk factors for back pain among workers in the construction industry. Participatory ergonomic initiatives increase the success of interventions aimed at reducing physical excessive exposures.

The objectives are in two phases to; 1) determine which work-tasks in selected job-groups involve the highest load of the back and shoulders during a normal working day (using EMG, Actigraphs, Video). 2) investigate whether a participatory intervention can reduce physical workloads, drawing on information from objective measurements from phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Full time construction workers who are member of a labor union and can read and understand Danish.
* The type of work must include manual work that involves lifting

Exclusion Criteria:

* life-threatening diseases
* pregnancy
* hypertension >160/100 mmHg
* unable to participate in the measurements

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Excessive physical load | change from baseline to 3 months follow-up
  The primary outcome of the present study is the change from baseline to follow-up in frequency of events with excessive physical load

SECONDARY OUTCOMES:
Pain intensity (0-10) | change from baseline to 3 months follow-up
  Change in "low back pain intensity during the last week" from baseline to follow-up. A horizontally oriented modified VAS scale will be used with 11 points from 0 to 10.
WAI questionnaire | change from baseline to 3 months follow-up
  Work Ability Index (Ilmarinen et al)
Self-efficacy Questionnaire | change from baseline to 3 months follow-up
  Self-efficacy to improve the physical work environment

OTHER OUTCOMES:
Social Capital questionnaire | change from baseline to 3 months follow-up
  Social Capital within work teams, between work teams, and between teams and their leaders Reference for questionnaire: http://www.ncbi.nlm.nih.gov/pubmed/26261190

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Study Director — National Research Centre for the Working Environment, Denmark
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

REFERENCES:
- [Derived] Brandt M, Madeleine P, Samani A, Ajslev JZ, Jakobsen MD, Sundstrup E, Andersen LL. Effects of a Participatory Ergonomics Intervention With Wearable Technical Measurements of Physical Workload in the Construction Industry: Cluster Randomized Controlled Trial. J Med Internet Res. 2018 Dec 19;20(12):e10272. doi: 10.2196/10272. PMID 30567694
- [Derived] Brandt M, Madeleine P, Ajslev JZ, Jakobsen MD, Samani A, Sundstrup E, Kines P, Andersen LL. Participatory intervention with objectively measured physical risk factors for musculoskeletal disorders in the construction industry: study protocol for a cluster randomized controlled trial. BMC Musculoskelet Disord. 2015 Oct 16;16:302. doi: 10.1186/s12891-015-0758-0. PMID 26474867